CLINICAL TRIAL: NCT04967599
Title: Alcohol Metabolism and Disease Risk in Asians: Examining the Impact of Personalized Phenotypic/Genotypic Feedback and Motivational Processes on Early Drinking Trajectories
Brief Title: Alcohol Metabolism and Disease Risk in Asians
Acronym: R21AA28365
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Susan Luczak, Professor (Research), University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-20-00814
Record Dates: First submitted 2021-06-29; First posted 2021-07-19 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Genes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (CONTROL) (No Intervention): Participants do not receive PHEN or GENE.
- Phenotype Feedback (PHEN) (Experimental): Participants receive the PHEN intervention.
  Interventions: Behavioral: Phenotype Feedback Intervention
- Phenotype and Genotype Feedback (PHEN+GENE) (Experimental): Participants receive the PHEN and GENE interventions.
  Interventions: Behavioral: Phenotype Feedback Intervention; Behavioral: Genotype Feedback Intervention

INTERVENTIONS:
Behavioral: Phenotype Feedback Intervention — Online session providing information on health-related risk associated with alcohol consumption and alcohol metabolism gene variations plus personalized feedback on flushing phenotype and associated risks.
  Other Names: PHEN
  Arms: Phenotype Feedback (PHEN); Phenotype and Genotype Feedback (PHEN+GENE)
Behavioral: Genotype Feedback Intervention — Online session providing personalized feedback on alcohol metabolism genotypes and associated health-related risks.
  Other Names: GENE
  Arms: Phenotype and Genotype Feedback (PHEN+GENE)

SUMMARY:
The primary pathway of alcohol metabolism involves two main enzymes, alcohol and aldehyde dehydrogenase. Several genes that encode these enzymes have variants that alter the rate of alcohol metabolism and increase levels of acetaldehyde. The variant ALDH2*2 allele is associated with the flushing response (i.e., Asian glow) and is found almost exclusively in individuals of east Asian descent. Although having variant ALDH2 alleles is protective against heavy drinking and alcohol use disorders, for those who do drink, these variants also are associated with elevations in risk for several health problems. The premise of this study is that we can affect early drinking behavior through personalized communication about these health-related risks.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be of Asian heritage (i.e. Chinese/Taiwanese, Japanese, Korean, Vietnamese).
* About half of the sample will be incoming first-year undergraduates
* About half of the sample will be current undergraduates who self-report having flushed when they first started drinking alcohol

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Luczak, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be uploaded to the National Institute of Mental Health Data Archive.
Time Frame: Data will be shared no later than 2 years after the project end date.
Access Criteria: De-identified data will be available to eligible researchers, and summary information will be available to the public.
URL: https://nda.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited July to October 2021 as a college student sample in Los Angeles
Pre-assignment Details: All 360 participants were assigned to a group.
Period: Overall Study
Arm/Group | Control (CONTROL) | Phenotype Feedback (PHEN) | Phenotype and Genotype Feedback (PHEN+GENE)
Started | 120 | 120 | 120
Completed | 85 | 101 | 97
Not Completed | 35 | 19 | 23
Not completed — Lost to Follow-up | 35 | 19 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (CONTROL) | Phenotype Feedback (PHEN) | Phenotype and Genotype Feedback (PHEN+GENE) | Total
Number analyzed (Participants) | 120 | 120 | 120 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.7 (1.1) | 19.1 (1.3) | 18.6 (1.2) | 18.8 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 68 | 74 | 208
  Male | 54 | 52 | 46 | 152
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 115 | 111 | 112 | 338
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 5 | 9 | 8 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 120 | 120 | 120 | 360

OUTCOME MEASURES:

1. Primary Outcome: Peak Number of Alcohol Drinks Consumed in a Day
Description: Drinking quantity (i.e. total number of alcoholic drinks) consumed on heaviest drinking day
Time Frame: Baseline through 10-months post-intervention (which occurred on 1 day)
Population: 360 participants were in the baseline assessment, 280 had this outcome in the 10-month follow-up assessment
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Control (CONTROL) | Phenotype Feedback (PHEN) | Phenotype and Genotype Feedback (PHEN+GENE)
Number analyzed (Participants) | 120 | 120 | 120
drinks
  Baseline | 3.7 (3.5) | 4.2 (4.1) | 3.4 (3.0)
  10-month follow-up: number analyzed (Participants) | 85 | 99 | 96
  10-month follow-up | 3.0 (2.9) | 2.8 (2.7) | 3.2 (3.5)
Statistical Analysis 1: Comparison: Control (CONTROL) vs Phenotype Feedback (PHEN) vs Phenotype and Genotype Feedback (PHEN+GENE); Test type: Superiority; p = .81, Kruskal-Wallis

2. Secondary Outcome: Number of Drinking Days
Description: Number of days consumed alcohol in the past month
Time Frame: Baseline through 10-months post-intervention (which occurred on 1 day)
Population: 360 participants were in the baseline assessment, 279 of whom reported this variable in the 10-month follow-up assessment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control (CONTROL) | Phenotype Feedback (PHEN) | Phenotype and Genotype Feedback (PHEN+GENE)
Number analyzed (Participants) | 120 | 120 | 120
days
  Baseline | 2.4 (1.8) | 2.3 (1.8) | 2.3 (1.8)
  10-month follow-up: number analyzed (Participants) | 85 | 99 | 95
  10-month follow-up | 2.3 (1.9) | 2.0 (1.8) | 2.2 (1.8)
Statistical Analysis 1: Comparison: Control (CONTROL) vs Phenotype Feedback (PHEN) vs Phenotype and Genotype Feedback (PHEN+GENE); Test type: Superiority; p = .46, Kruskal-Wallis

3. Secondary Outcome: Number of Alcoholic Drinks Consumed on Weekend
Description: Alcohol quantity (total number of drinks) consumed on a typical drinking weekend
Time Frame: Baseline through 10-months post-intervention (which occurred on 1 day)
Population: 360 participants were in the baseline assessment, 269 of whom reported on this variable in the 10-month follow-up assessment
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Control (CONTROL) | Phenotype Feedback (PHEN) | Phenotype and Genotype Feedback (PHEN+GENE)
Number analyzed (Participants) | 120 | 120 | 120
drinks
  Baseline | 2.7 (4.2) | 3.1 (4.4) | 2.7 (3.6)
  10-month follow-up: number analyzed (Participants) | 82 | 93 | 94
  10-month follow-up | 2.1 (3.8) | 1.9 (3.0) | 2.7 (4.2)
Statistical Analysis 1: Comparison: Control (CONTROL) vs Phenotype Feedback (PHEN) vs Phenotype and Genotype Feedback (PHEN+GENE); Test type: Superiority; p = .49, Kruskal-Wallis

4. Secondary Outcome: Number of Alcoholic Drinks Consumed Weekly
Description: Total quantity (i.e. number of drinks) of alcohol consumed in a typical drinking week
Time Frame: Baseline through 10-months post-intervention (which occurred on 1 day)
Population: 360 participants were in the baseline assessment, 269 of whom reported this variable in the 10-month follow-up
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Control (CONTROL) | Phenotype Feedback (PHEN) | Phenotype and Genotype Feedback (PHEN+GENE)
Number analyzed (Participants) | 120 | 120 | 120
drinks
  Baseline | 3.2 (4.6) | 4.0 (5.6) | 2.9 (4.1)
  10-month follow-up: number analyzed (Participants) | 82 | 93 | 94
  10-month follow-up | 2.8 (5.8) | 2.2 (3.4) | 2.7 (4.2)
Statistical Analysis 1: Comparison: Control (CONTROL) vs Phenotype Feedback (PHEN) vs Phenotype and Genotype Feedback (PHEN+GENE); Test type: Superiority; p = .59, Kruskal-Wallis

5. Secondary Outcome: Number of Participants Identified as Non-drinkers
Description: Number of Participants Identified as Non-drinkers (i.e. have not had alcohol beyond small sips or tastes)
Time Frame: Baseline through 10-months post-intervention (which occurred on 1 day)
Population: 360 participants were in the baseline assessment, 280 of whom reported on this variable in the 10-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Control (CONTROL) | Phenotype Feedback (PHEN) | Phenotype and Genotype Feedback (PHEN+GENE)
Number analyzed (Participants) | 120 | 120 | 120
Participants
  Baseline | 14 | 15 | 16
  10-month follow-up: number analyzed (Participants) | 85 | 99 | 96
  10-month follow-up | 4 | 9 | 4
Statistical Analysis 1: Comparison: Control (CONTROL) vs Phenotype Feedback (PHEN) vs Phenotype and Genotype Feedback (PHEN+GENE); Test type: Superiority; p = .29, Fisher Exact

6. Secondary Outcome: Alcohol Flush Cure Use Rate
Description: Proportion of time used a product to reduce flushing when drinking alcohol
Time Frame: Baseline through 10-months post-intervention (which occurred on 1 day)
Population: 311 participants in the baseline assessment and 220 in the 10-month follow-up assessment were current drinkers and could have used a flush cure (i.e. taken a substance to reduce flushing when drinking alcohol)
Measure: Count of Participants; unit: Participants
Arm/Group | Control (CONTROL) | Phenotype Feedback (PHEN) | Phenotype and Genotype Feedback (PHEN+GENE)
Number analyzed (Participants) | 107 | 101 | 103
Participants
  Baseline: Some of the time used a flush cure | 7 | 6 | 3
  Baseline: Almost never/never used a flush cure | 97 | 91 | 94
  Baseline: Half of the time or more used a flush cure | 3 | 4 | 6
  10-month follow-up: number analyzed (Participants) | 68 | 74 | 78
  10-month follow-up: Some of the time used a flush cure | 5 | 2 | 2
  10-month follow-up: Almost never/never used a flush cure | 61 | 67 | 73
  10-month follow-up: Half of the time or more used a flush cure | 2 | 5 | 3
Statistical Analysis 1: Comparison: Control (CONTROL) vs Phenotype Feedback (PHEN) vs Phenotype and Genotype Feedback (PHEN+GENE); Test type: Superiority; p = .49, Fisher Exact

ADVERSE EVENTS:
Time Frame: This study provided a brief informational online intervention session to participants so no information on adverse medical event data were obtained.
Description: This study provided a brief informational online intervention session to participants so no information on adverse medical event data were obtained.
Arm/Group | Control (CONTROL) | Phenotype Feedback (PHEN) | Phenotype and Genotype Feedback (PHEN+GENE)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04967599/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04967599/ICF_001.pdf